CLINICAL TRIAL: NCT06448377
Title: Initiation of Airway Code: the Role of the Airway Team in Unexpected Difficult Airways
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-25
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-06

CONDITIONS: Unexpected Difficult Airway; Intubation;Difficult; Airway Management
Keywords: airway management; anesthesia; intubation; difficult airway
MeSH Terms: interventions — Intubation, Intratracheal; Laryngoscopy; Bro protein, Drosophila

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Airway Team Group: In this group, the intervention time and methods used by the airway team will be evaluated in patients who have been called for airway assistance.
  Interventions: Procedure: Videolaryngoscopy; Procedure: FOB; Procedure: FOB+Aintree; Procedure: Classic intubation with laryngoscopy; Procedure: Others
- Control Group: In this group, anesthesiologists' feedback on difficult airway cases will be received.
  Interventions: Procedure: Videolaryngoscopy; Procedure: FOB; Procedure: FOB+Aintree; Procedure: Classic intubation with laryngoscopy; Procedure: Others

INTERVENTIONS:
Procedure: Videolaryngoscopy — Situations in which the practitioner performs endotracheal intubation using a videolaryngoscope during airway intervention will be included in this group.
Procedure: FOB — Situations in which the practitioner performs endotracheal intubation using a fiberoptic bronchoscope during airway intervention will be included in this group.
  Other Names: endotracheal intubation with fiberoptic bronchoscope
Procedure: FOB+Aintree — Situations in which the practitioner performs endotracheal intubation using a Fiberoptic intubation via LMA with aintree catheter during airway intervention will be included in this group.
  Other Names: Fiberoptic intubation via LMA with aintree catheter
Procedure: Classic intubation with laryngoscopy — Situations in which the practitioner performs endotracheal intubation using a macintosh laryngoscope during airway intervention will be included in this group.
Procedure: Others — Cases in which intubation cannot be performed, those who are awakened from anesthesia, or those in whom a surgical method is used for airway access will be included in this group.

SUMMARY:
The aim of our study is to observationally examine our unexpected difficult airway incidence and intervention times. In addition, it is aimed to discuss the clinical effect of a team specialized in airway intervention intervening in cases by call on the success of airway intervention. In this discussion, it is aimed to use the opinion-opposition method.

DETAILED DESCRIPTION:
Initiation of Airway Code: The Role of the Airway Team in Unexpected Difficult Airways

The incidence of difficult airway is approximately 1 in 1000 cases and poses a significant perioperative risk to patients. Various classifications, guidelines, and approaches have been developed to identify patients with difficult airways. However, even the most well-known classifications are not 100% successful in predicting difficult airways. Consequently, some unexpected difficult airway cases are encountered, and their management continues to be a subject of new research in the literature.

In situations involving difficult airways, having the same team respond to every case may pose a potential obstacle to the distribution of experience and responsibilities among other clinical staff. However, it is undeniable that experienced anesthetists are more successful in airway management, and the importance of airway-related training cannot be overstated. Similar to the code blue protocol used during cardiac arrests, the intervention of a trained external team in crisis situations, utilizing familiar equipment and applying data from previous cases for quality improvement, can provide significant benefits in airway management akin to those seen in cardiac arrests. This approach could also potentially enhance patient safety in internal medicine and surgical wards, as well as in certain intensive care units, where familiarity with airway management is limited.

This study aims to discuss the positive and negative impacts of the airway teams intervention in unexpected difficult airway situations within the operating room, using a pro-con debate method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be operated under general anesthesia at Kocaeli City Hospital or who require perioperative endotracheal intubation will be included in our study.
2. Operations performed within the study time period will be taken
3. Patients whose anesthesiologists call for help for difficult airway will be included in the study.
4. Patients between the ages of 18-65 will be included in the study.

Exclusion Criteria:

- 1. Expected difficult airway patients (mallampati 3-4) and other patients with high difficult airway scores will not be included in the study.

2. Patients with difficult airway conditions but who will be awakened by giving up endotracheal intubation will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unexpected difficult airway patients will be included in our study. These patients should need perioperative endotracheal intubation without signs of difficult airway in their airway evaluation scores, and the patients should be intervened by the anesthesiologists themselves or the airway team.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Successful endotracheal intubation rate in difficult airway | During the intraoperative period of difficult intubation case
  The primary outcome of our study is the rate( in percent) of complication-free and successful endotracheal intubation performed by specialists or the airway team in unexpected difficult airway cases.

SECONDARY OUTCOMES:
The response time of the airway team to the case and the tools they used | During the intraoperative period of difficult intubation case
  In this section, the interventions performed by the airway team will be compared with the control group. The duration( time in minutes) of the intervention and the different airway tools used will be compared numerically.
airway intervention equipment | During the intraoperative period of difficult intubation case
  To determine the most commonly used assistive devices (type) in airway intervention and to compare their frequencies ( in percent) in two different defined groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YUKSEK, Md, Principal Investigator — Kocaeli Cith Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study participants can be requested from Kocaeli Provincial Health Directorate with an appropriate letter. It is unauthorized for responsible researchers to distribute these data.

REFERENCES:
- [Background] Pandian V, Ghazi TU, He MQ, Isak E, Saleem A, Semler LR, Capellari EC, Brenner MJ. Multidisciplinary Difficult Airway Team Characteristics, Airway Securement Success, and Clinical Outcomes: A Systematic Review. Ann Otol Rhinol Laryngol. 2023 Aug;132(8):938-954. doi: 10.1177/00034894221123124. Epub 2022 Oct 2. PMID 36189709
- [Background] Karamchandani K, Wheelwright J, Yang AL, Westphal ND, Khanna AK, Myatra SN. Emergency Airway Management Outside the Operating Room: Current Evidence and Management Strategies. Anesth Analg. 2021 Sep 1;133(3):648-662. doi: 10.1213/ANE.0000000000005644. PMID 34153007
- [Background] Penketh J, Nolan JP. Airway management during cardiac arrest. Curr Opin Crit Care. 2023 Jun 1;29(3):175-180. doi: 10.1097/MCC.0000000000001033. Epub 2023 Mar 28. PMID 37078613
- [Background] Mark LJ, Herzer KR, Cover R, Pandian V, Bhatti NI, Berkow LC, Haut ER, Hillel AT, Miller CR, Feller-Kopman DJ, Schiavi AJ, Xie YJ, Lim C, Holzmueller C, Ahmad M, Thomas P, Flint PW, Mirski MA. Difficult airway response team: a novel quality improvement program for managing hospital-wide airway emergencies. Anesth Analg. 2015 Jul;121(1):127-139. doi: 10.1213/ANE.0000000000000691. PMID 26086513
- [Background] Koh W, Kim H, Kim K, Ro YJ, Yang HS. Encountering unexpected difficult airway: relationship with the intubation difficulty scale. Korean J Anesthesiol. 2016 Jun;69(3):244-9. doi: 10.4097/kjae.2016.69.3.244. Epub 2016 Jun 1. PMID 27274369